CLINICAL TRIAL: NCT01675674
Title: Unrecognized Mucopolysaccharidosis I, II, IVA, and VI in the Pediatric Rheumatology Population
Brief Title: Study to Detect Unrecognized Mucopolysaccharidosis in Children Visiting Rheumatology, Hand or Skeletal Dysplasia Clinics
Status: Terminated | Type: Observational
Why Stopped: Funding withdrawn due to insufficient enrollment rate
Sponsor: National MPS Society (Other)
Collaborators: MediResource Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: RHE-001
Record Dates: First submitted 2012-08-23; First posted 2012-08-30 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Mucopolysaccharidoses; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI
Keywords: Mucopolysaccharidoses; Prevalence; Pediatric; Rheumatology; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI
MeSH Terms: conditions — Mucopolysaccharidoses; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dried blood spot test for MPS: For the prospective study, subjects will be drawn from all children (aged 6 months to 18 years) with a history of presenting to selected clinics (pediatric rheumatology, pediatric hand, or skeletal dysplasia clinic), with at least ONE "highly suspicious" symptom or at least TWO "less suspicious" symptoms that may be indicative of an MPS disorder (see inclusion criteria).
  For the retrospective chart review, subjects will be drawn from all children who were 6 months to 18 years of age at the time of first presentation to selected clinics (pediatric rheumatology, pediatric hand, or skeletal dysplasia clinic), with at least ONE "highly suspicious" symptom or at least TWO "less suspicious" symptoms that may be indicative of an MPS disorder (see inclusion criteria).
  Interventions: Other: Dried blood spot test for MPS

INTERVENTIONS:
Other: Dried blood spot test for MPS — The dried blood spot test uses a few drops of blood on filter paper to screen for mucopolysaccharidoses (MPS I, MPS II, MPS IVA and MPS VI in this study).
  Other Names: DBS testing

SUMMARY:
This study is being done to learn how many children and young adults who come to pediatric rheumatology clinics may have mucopolysaccharidosis (MPS). The study tests for 4 of the types of MPS: I, II, IVA, and VI. This can help researchers decide whether to create a screening program for MPS at pediatric rheumatology clinics. This study is being done in rheumatology clinics because the first symptoms of MPS are often joint problems such as stiff joints, and rheumatologists may be the first doctors that a patient with MPS visits. The study will also evaluate the utility of dried blood spot testing for MPS.

DETAILED DESCRIPTION:
MPS, or mucopolysaccharidosis (mew-co-paw-lee-sack-a-rid-o-sis), disorders are a group of rare inherited diseases that affect about 1 in every 25,000 people in the United States. There are 7 MPS disorders: MPS I (Hurler, Hurler-Scheie, and Scheie syndromes), II (Hunter syndrome), III (Sanfilippo syndrome), IV (Morquio syndrome), VI (Maroteaux-Lamy syndrome), VII (Sly syndrome), and IX (no other name). In people who have MPS, the body cannot break down certain materials in the body's cells. These materials then build up in the cells, causing problems such as stiff joints, misshapen bones, curled hands and reduced hand function, frequent ear infections, vision and hearing problems, "thickened" facial features, and heart problems. Getting access to diagnosis and treatment can help make MPS easier to manage; but unfortunately, people with MPS may go undiagnosed for many years.

This study is being done to learn how many children and young adults who come to pediatric rheumatology clinics may have mucopolysaccharidosis (MPS). The study tests for 4 of the types of MPS: I, II, IVA, and VI. This can help researchers decide whether to create a screening program for MPS at pediatric rheumatology clinics. This study is being done in rheumatology clinics because the first symptoms of MPS are often joint problems such as stiff joints, and rheumatologists may be the first doctors that a patient with MPS visits.

The study will use dried blood spot (DBS) testing to screen for these types of MPS. It will also use a survey to evaluate the utility and convenience of dried blood spot testing for MPS.

ELIGIBILITY:
Inclusion Criteria:

1. History of presenting to the pediatric rheumatology, pediatric hand, or skeletal dysplasia clinic with at least ONE "highly suspicious" symptom or at least TWO "less suspicious" symptoms that may be indicative of an MPS disorder (see below):

   Highly suspicious symptoms:
   * characteristic facial features
   * hearing loss
   * corneal clouding
   * cardiac manifestations
   * dysostosis multiplex
   * hepatosplenomegaly
   * spinal cord compression
   * hydrocephalus
   * carpal tunnel syndrome
   * delayed mental development or regression in mental development

   Less suspicious symptoms:
   * short stature
   * extensive Mongolian spots
   * sleep apnea
   * copious nasal discharge
   * recurrent otitis media, ear fluid that will not drain, or the presence of ear tubes
   * frequent upper respiratory tract infections
   * joint stiffness or limited range of motion
   * hand problems (Claw hands or reduced hand function)
   * hernia (inguinal or umbilical)
   * abnormally shaped teeth
   * dental cysts
   * tooth abscess
2. Age of at least 6 months.
3. Age under 18 years at time of initial clinic presentation.
4. Written, signed, and dated informed consent obtained from the subject (if 18 years of age) or the subject's parents (if under 18). Written, dated, and signed assent from children is also required at some centers.

Exclusion Criteria:

1. Under 6 months of age.
2. Over 18 years of age at initial clinic presentation.
3. Patients who have had confirmation of an MPS disorder by biochemical analysis and/or by molecular biology.
4. Patients for whom MPS enzyme activity tests (i.e., enzyme levels tested in fibroblasts, leukocytes, serum, or blood spots) have already been performed, and for which the result was normal. (Patients who have been screened for MPS through urinary GAG and tested normal will not be excluded from the study.)
5. Written informed consent not available.
6. Subject unwilling or unable to provide the necessary blood spot for analysis.
7. Any other condition that would, in the opinion of the investigator, interfere with the participant's ability to provide informed consent, comply with study instructions, or possibly confound interpretation of study results.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For the prospective study, subjects will be drawn from all children (aged 6 months to 18 years) with a history of presenting to selected clinics (pediatric rheumatology, pediatric hand, or skeletal dysplasia clinic), with at least ONE "highly suspicious" symptom or at least TWO "less suspicious" symptoms that may be indicative of an MPS disorder (see inclusion criteria).
  For the retrospective chart review, subjects will be drawn from all children who were 6 months to 18 years of age at the time of first presentation to selected clinics (pediatric rheumatology, pediatric hand, or skeletal dysplasia clinic), with at least ONE "highly suspicious" symptom or at least TWO "less suspicious" symptoms that may be indicative of an MPS disorder (see inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of previously unrecognized MPS I, II, IVA, and VI in children presenting to pediatric rheumatology, hand, or skeletal dysplasia clinics | At study completion (approximately 18 months after the beginning of the study)
  Each patient is screened for MPS I, II, IVA, and VI after enrolling in the study. The results for all patients will be pooled when the study is completed (expected completion approx. 18 months after the study begins).

SECONDARY OUTCOMES:
Utility of DBS testing to screen for MPS in pediatric patients | At study completion (approximately 18 months after the beginning of the study)
  For the secondary endpoint (utility of DBS testing), the following data will be collected: ease of taking and sending the DBS sample; number of errors of sample taking; adverse events (if any) associated with blood sampling by finger prick or venipuncture (for subjects over one year of age; choose whichever method is most convenient) or heel prick (for subjects under one year of age); and comfort of patients and/or their parents with the test.
  Study personnel who performed DBS testing will also be asked to complete a brief survey about the utility of DBS testing.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas JA Lehman, MD, Principal Investigator — Chief, Division of Pediatric Rheumatology, Hospital for Special Surgery; Professor of Clinical Pediatrics, Cornell University
Locations (2):
- United States (2):
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York

REFERENCES:
- [Background] Cimaz R, Coppa GV, Kone-Paut I, Link B, Pastores GM, Elorduy MR, Spencer C, Thorne C, Wulffraat N, Manger B. Joint contractures in the absence of inflammation may indicate mucopolysaccharidosis. Pediatr Rheumatol Online J. 2009 Oct 23;7:18. doi: 10.1186/1546-0096-7-18. PMID 19852785
- [Background] Baehner F, Schmiedeskamp C, Krummenauer F, Miebach E, Bajbouj M, Whybra C, Kohlschutter A, Kampmann C, Beck M. Cumulative incidence rates of the mucopolysaccharidoses in Germany. J Inherit Metab Dis. 2005;28(6):1011-7. doi: 10.1007/s10545-005-0112-z. PMID 16435194
- [Background] Lin HY, Lin SP, Chuang CK, Niu DM, Chen MR, Tsai FJ, Chao MC, Chiu PC, Lin SJ, Tsai LP, Hwu WL, Lin JL. Incidence of the mucopolysaccharidoses in Taiwan, 1984-2004. Am J Med Genet A. 2009 May;149A(5):960-4. doi: 10.1002/ajmg.a.32781. PMID 19396827
- [Background] Malm G, Lund AM, Mansson JE, Heiberg A. Mucopolysaccharidoses in the Scandinavian countries: incidence and prevalence. Acta Paediatr. 2008 Nov;97(11):1577-81. doi: 10.1111/j.1651-2227.2008.00965.x. Epub 2008 Aug 4. PMID 18681890
- [Background] Moore D, Connock MJ, Wraith E, Lavery C. The prevalence of and survival in Mucopolysaccharidosis I: Hurler, Hurler-Scheie and Scheie syndromes in the UK. Orphanet J Rare Dis. 2008 Sep 16;3:24. doi: 10.1186/1750-1172-3-24. PMID 18796143
- [Background] Murphy AM, Lambert D, Treacy EP, O'Meara A, Lynch SA. Incidence and prevalence of mucopolysaccharidosis type 1 in the Irish republic. Arch Dis Child. 2009 Jan;94(1):52-4. doi: 10.1136/adc.2007.135772. Epub 2008 May 7. PMID 18463126
- [Background] Nelson J, Crowhurst J, Carey B, Greed L. Incidence of the mucopolysaccharidoses in Western Australia. Am J Med Genet A. 2003 Dec 15;123A(3):310-3. doi: 10.1002/ajmg.a.20314. PMID 14608657
- [Background] Poorthuis BJ, Wevers RA, Kleijer WJ, Groener JE, de Jong JG, van Weely S, Niezen-Koning KE, van Diggelen OP. The frequency of lysosomal storage diseases in The Netherlands. Hum Genet. 1999 Jul-Aug;105(1-2):151-6. doi: 10.1007/s004399900075. PMID 10480370
- [Background] Verity C, Winstone AM, Stellitano L, Will R, Nicoll A. The epidemiology of progressive intellectual and neurological deterioration in childhood. Arch Dis Child. 2010 May;95(5):361-4. doi: 10.1136/adc.2009.173419. Epub 2009 Nov 29. PMID 19948513
- [Background] Giugliani R, Harmatz P, Wraith JE. Management guidelines for mucopolysaccharidosis VI. Pediatrics. 2007 Aug;120(2):405-18. doi: 10.1542/peds.2006-2184. PMID 17671068
- [Background] Muenzer J, Wraith JE, Clarke LA; International Consensus Panel on Management and Treatment of Mucopolysaccharidosis I. Mucopolysaccharidosis I: management and treatment guidelines. Pediatrics. 2009 Jan;123(1):19-29. doi: 10.1542/peds.2008-0416. PMID 19117856
- [Background] Muenzer J, Beck M, Eng CM, Escolar ML, Giugliani R, Guffon NH, Harmatz P, Kamin W, Kampmann C, Koseoglu ST, Link B, Martin RA, Molter DW, Munoz Rojas MV, Ogilvie JW, Parini R, Ramaswami U, Scarpa M, Schwartz IV, Wood RE, Wraith E. Multidisciplinary management of Hunter syndrome. Pediatrics. 2009 Dec;124(6):e1228-39. doi: 10.1542/peds.2008-0999. Epub 2009 Nov 9. PMID 19901005
- [Background] Aldenhoven M, de Koning TJ, Verheijen FW, Prinsen BH, Wijburg FA, van der Ploeg AT, de Sain-van der Velden MG, Boelens J. Dried blood spot analysis: an easy and reliable tool to monitor the biochemical effect of hematopoietic stem cell transplantation in hurler syndrome patients. Biol Blood Marrow Transplant. 2010 May;16(5):701-4. doi: 10.1016/j.bbmt.2010.01.006. Epub 2010 Jan 21. PMID 20096360
- [Background] Chamoles NA, Blanco MB, Gaggioli D, Casentini C. Hurler-like phenotype: enzymatic diagnosis in dried blood spots on filter paper. Clin Chem. 2001 Dec;47(12):2098-102. PMID 11719472
- [Background] Chamoles NA, Blanco M, Gaggioli D. Diagnosis of alpha-L-iduronidase deficiency in dried blood spots on filter paper: the possibility of newborn diagnosis. Clin Chem. 2001 Apr;47(4):780-1. No abstract available. PMID 11274042
- [Background] Gelb MH, Turecek F, Scott CR, Chamoles NA. Direct multiplex assay of enzymes in dried blood spots by tandem mass spectrometry for the newborn screening of lysosomal storage disorders. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):397-404. doi: 10.1007/s10545-006-0265-4. PMID 16763908
- [Background] Wang D, Eadala B, Sadilek M, Chamoles NA, Turecek F, Scott CR, Gelb MH. Tandem mass spectrometric analysis of dried blood spots for screening of mucopolysaccharidosis I in newborns. Clin Chem. 2005 May;51(5):898-900. doi: 10.1373/clinchem.2004.047167. Epub 2005 Feb 3. No abstract available. PMID 15695324
- [Background] Blanchard S, Sadilek M, Scott CR, Turecek F, Gelb MH. Tandem mass spectrometry for the direct assay of lysosomal enzymes in dried blood spots: application to screening newborns for mucopolysaccharidosis I. Clin Chem. 2008 Dec;54(12):2067-70. doi: 10.1373/clinchem.2008.115410. PMID 19042989
- [Background] Dean CJ, Bockmann MR, Hopwood JJ, Brooks DA, Meikle PJ. Detection of mucopolysaccharidosis type II by measurement of iduronate-2-sulfatase in dried blood spots and plasma samples. Clin Chem. 2006 Apr;52(4):643-9. doi: 10.1373/clinchem.2005.061838. Epub 2006 Feb 23. PMID 16497940
- [Background] Wang D, Wood T, Sadilek M, Scott CR, Turecek F, Gelb MH. Tandem mass spectrometry for the direct assay of enzymes in dried blood spots: application to newborn screening for mucopolysaccharidosis II (Hunter disease). Clin Chem. 2007 Jan;53(1):137-40. doi: 10.1373/clinchem.2006.077263. Epub 2006 Nov 2. PMID 17082248
- [Background] Wolfe BJ, Blanchard S, Sadilek M, Scott CR, Turecek F, Gelb MH. Tandem mass spectrometry for the direct assay of lysosomal enzymes in dried blood spots: application to screening newborns for mucopolysaccharidosis II (Hunter Syndrome). Anal Chem. 2011 Feb 1;83(3):1152-6. doi: 10.1021/ac102777s. Epub 2010 Dec 30. PMID 21192662
- [Background] Parkinson-Lawrence EJ, Muller VJ, Hopwood JJ, Brooks DA. N-acetylgalactosamine-6-sulfatase protein detection in MPS IVA patient and unaffected control samples. Clin Chim Acta. 2007 Feb;377(1-2):88-91. doi: 10.1016/j.cca.2006.08.030. Epub 2006 Sep 1. PMID 17027703
- [Background] Hein LK, Meikle PJ, Dean CJ, Bockmann MR, Auclair D, Hopwood JJ, Brooks DA. Development of an assay for the detection of mucopolysaccharidosis type VI patients using dried blood-spots. Clin Chim Acta. 2005 Mar;353(1-2):67-74. doi: 10.1016/j.cccn.2004.10.009. PMID 15698592
- [Background] Duffey TA, Sadilek M, Scott CR, Turecek F, Gelb MH. Tandem mass spectrometry for the direct assay of lysosomal enzymes in dried blood spots: application to screening newborns for mucopolysaccharidosis VI (Maroteaux-Lamy syndrome). Anal Chem. 2010 Nov 15;82(22):9587-91. doi: 10.1021/ac102090v. Epub 2010 Oct 20. PMID 20961069
- [Background] Ashrafi MR, Shabanian R, Mohammadi M, Kavusi S. Extensive Mongolian spots: a clinical sign merits special attention. Pediatr Neurol. 2006 Feb;34(2):143-5. doi: 10.1016/j.pediatrneurol.2005.07.010. PMID 16458829
- [Background] Ochiai T, Suzuki Y, Kato T, Shichino H, Chin M, Mugishima H, Orii T. Natural history of extensive Mongolian spots in mucopolysaccharidosis type II (Hunter syndrome): a survey among 52 Japanese patients. J Eur Acad Dermatol Venereol. 2007 Sep;21(8):1082-5. doi: 10.1111/j.1468-3083.2007.02203.x. PMID 17714129
- [Background] Wraith JE, Scarpa M, Beck M, Bodamer OA, De Meirleir L, Guffon N, Meldgaard Lund A, Malm G, Van der Ploeg AT, Zeman J. Mucopolysaccharidosis type II (Hunter syndrome): a clinical review and recommendations for treatment in the era of enzyme replacement therapy. Eur J Pediatr. 2008 Mar;167(3):267-77. doi: 10.1007/s00431-007-0635-4. Epub 2007 Nov 23. PMID 18038146
- [Background] Hendley JO. Clinical practice. Otitis media. N Engl J Med. 2002 Oct 10;347(15):1169-74. doi: 10.1056/NEJMcp010944. No abstract available. PMID 12374878
- [Background] Rovers MM, Balemans WA, Sanders EA, van der Ent CK, Zielhuis GA, Schilder AG. Persistence of upper respiratory tract infections in a cohort followed from childhood to adulthood. Fam Pract. 2006 Jun;23(3):286-90. doi: 10.1093/fampra/cml001. Epub 2006 Mar 3. PMID 16517546
- [Background] Tomatsu S, Nishioka T, Montano AM, Gutierrez MA, Pena OS, Orii KO, Sly WS, Yamaguchi S, Orii T, Paschke E, Kircher SG, Noguchi A. Mucopolysaccharidosis IVA: identification of mutations and methylation study in GALNS gene. J Med Genet. 2004 Jul;41(7):e98. doi: 10.1136/jmg.2003.018010. No abstract available. PMID 15235041